CLINICAL TRIAL: NCT02156921
Title: Cost-effectiveness of Mobile App-guided Training in Extended Focused Assessment With Sonography for Trauma (eFAST): A Randomized Trial
Brief Title: App-guided Training in eFAST Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen Academy for Medical Education and Simulation (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Philip Mørkeberg Nilsson, Research Assistant, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H-3-2014-FSP17
Record Dates: First submitted 2014-05-27; First posted 2014-06-05 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Learning Outcome; Training Efficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Self-guided training without app-based training (written hand-outs)
- Intervention group (Active Comparator): Self-guided training with app-based training
  Interventions: Other: App-based training

INTERVENTIONS:
Other: App-based training
  Arms: Intervention group

SUMMARY:
This study aims to investigate the cost-effectiveness of app-based self-directed ultrasound training compared to self-directed training with written handouts on subsequent performance on simulated patient cases and theoretical cases.

ELIGIBILITY:
Inclusion Criteria:

* First year medical doctor
* Provided written informed consent

Exclusion Criteria:

* Prior practical ultrasonography experience such as performing independent ultrasonography scans, or participation in any post-graduate ultrasonography courses.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Video recording of ultrasound skills, rated by consultant radiologists. | Ratings are to be completed within three months of performance.
  The video-recordings of the technical performances are merged with the ultrasonography screen-recordings to one anonymized video-clip. These combined video-clips are rated with the OSAUS rating by two raters. The OSAUS scale (Objective Structured Assessment of Ultrasound Skills) is used for all performance assessments. The raters are consultant radiologists.
Cost-effectiveness of mobile app guided versus textbook guided training | September 2016

SECONDARY OUTCOMES:
Diagnostic accuracy | On site via checklist, evaluated on average one day after performance.
  Participants are given five videocases, to assess for eFAST verifiable pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Nilsson, Principal Investigator — Copenhagen Academy Of Medical Education And Simulation
Locations (1):
- Copenhagen Academy for Medical Education and Simulation, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No